CLINICAL TRIAL: NCT04102293
Title: Time Efficiency and Obturation Quality of Rotary Files Versus Manual Files in Pediatric Endodontics
Brief Title: Time Efficiency and Obturation Quality of Rotary Versus Manual in Primary Teeth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Reem Mahmoud Abdelkader Awad (Other)
Responsible Party: Sponsor-Investigator, Reem Mahmoud Abdelkader Awad, assistant lecturer, British University In Egypt
Organization: British University In Egypt (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PED19-2D
Record Dates: First submitted 2019-09-17; First posted 2019-09-25 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Endodontic Disease
Keywords: rotatry instrumentation
MeSH Terms: conditions — Dental Pulp Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Rotary instrumentation using MM files 1 (Experimental): Rotary instrumentation using MM files (IMD Inc, China), sizes 20-25-30 taper 0.4, length 16 mm, then obturation with Zinc oxide and Eugenol using Incremental filling Technique.
  Interventions: Procedure: NSK Endo motor Endomate
- Manual instrumentation using K-files 1 (Active Comparator): Manual instrumentation using K-files (Mani Inc, Tochigi, Japan), sizes 15-20-25-30-35 then obturation with Zinc oxide and Eugenol using Incremental filling Technique.
  Interventions: Procedure: manual K-files
- Rotary instrumentation using MM files 2 (Experimental): Rotary instrumentation using MM files (IMD Inc, China), sizes 20-25-30 taper 0.4, length 16 mm, then obturation with Zinc oxide and Eugenol using Disposable syringe technique.
  Interventions: Procedure: NSK Endo motor Endomate
- Manual instrumentation using K-files 2 (Active Comparator): Manual instrumentation using K-files (Mani Inc, Tochigi, Japan), sizes 15-20-25-30-35 then obturation with Zinc oxide and Eugenol using Disposable syringe technique
  Interventions: Procedure: manual K-files

INTERVENTIONS:
Procedure: NSK Endo motor Endomate — Rotary instrumenation used in pulp therapy
  Arms: Rotary instrumentation using MM files 1; Rotary instrumentation using MM files 2
Procedure: manual K-files — manual instrumentation used in pulp therapy
  Arms: Manual instrumentation using K-files 1; Manual instrumentation using K-files 2

SUMMARY:
The aim of this study is to evaluate the quality of obturation and the time efficiency of rotary versus manual instrumentation in roots of deciduous molars clinically where the:

* Primary objective Is to evaluate the time efficiency
* Secondary objective Is to evaluate the quality of obturation Clinical and radiographical follow up will be performed for 18 months to investigate the clinical and the radiographic success for the Conventional and Rotary groups.

DETAILED DESCRIPTION:
The study will be conducted in two parts as follows:

In-vitro part as a training part to practice, test the speed of the rotary system, followed by application clinically.

Obturation will be done using two different filling techniques:

* Incremental filling Technique
* Disposable syringe Technique.

Then the instrumentation time and the quality of obturation will be recorded.

The study will be conducted by recruiting patients from the Outpatient clinic of The Pediatric Dentistry and Dental Public Health department, Faculty of Dentistry, Ain Shams University:

ELIGIBILITY:
Inclusion Criteria:

-

Children included in the study should conform to the following criteria:

1. Patients between ages 4-7 years old with at least one mandibular vital or non-vital primary molar indicated for pulpectomy will be selected.
2. Absence of periapical or interadicular radiolucencies, inflammatory root resorption, sinus tract or gingival abscess.
3. No physiological root resorption.
4. The teeth should have enough coronal structure for full coverage Stainless-Steel crowns.

Exclusion Criteria:

* 1. Children who are extremely uncooperative and difficult to manage 2. Children suffering from any physically or mentally disability that will complicate the treatment: Special Health Care needs (SHCN) 3. Teeth of poor prognosis due to presence of an abscess or a sinus, mobility, advanced bone or root resorption or Non-Restorable teeth.

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 41 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Is to evaluate the time efficiency of the rotary mm files versus manual stainless steel k files in the pulpectomy of lower second primary molars affecting the positive behavior of the child | up to 18 months
  Time efficiency of instrumentation using rotary mm files specially designed for primary teeth versus manual stainless steel K-files in the pulpectomy of mandibular second primary molars, by clinical and radiographic evaluation for 18 months.
Is to evaluate and compare the quality of obturation using two different obturation techniques following instrumentation by rotary mm files and manual stainless steel k files instrumentation in another group | up to 18 months
  The quality of obturation using ZOE will be performed with either the incremental technique or the modified disposable syringe technique, following instrumentation by rotary and manual files, where the grading will be as : 1: overfilled, 2: underfilled 3: optimum filling.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams Univeristy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No